CLINICAL TRIAL: NCT02448498
Title: Strength Training Regimen for Normal Weight Diabetics
Acronym: STRONG-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Latha Palaniappan, MD, MS, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 32113
Record Dates: First submitted 2015-03-06; First posted 2015-05-19 (Estimated); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

ARMS (3):
- Strength Training Only (Experimental): Participants in the strength-training only group will take part in a 9-month exercise intervention at a local exercise facility. They will engage in strength training 3 days per week for approximately 60 minutes each exercise session.
  Interventions: Behavioral: Exercise Intervention
- Aerobic Training Only (Experimental): Participants in the aerobic training only group will take part in a 9-month exercise intervention at a local exercise facility. They will engage in aerobic training over 3 -5 days per week to achieve the targeted dose of 12 kcal/kg per week at a training intensity between 50-80% VO2 max.
  Interventions: Behavioral: Exercise Intervention
- Combination (Strength and Aerobic) Training (Experimental): Participants in the combination (strength and aerobic training) group will take part in a 9-month exercise intervention at a local exercise facility. They will engage aerobic training that will expend 10 kcal/kg/week in combination with strength-training, 3 days per week.
  Interventions: Behavioral: Exercise Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention

SUMMARY:
The Strength Training Regimen in Normal Weight Diabetics (STRONG-D) study will examine the effectiveness of different exercise regimen types in controlling diabetes for the normal weight type 2 diabetes population.

DETAILED DESCRIPTION:
In the STRONG-D study, participants are randomly assigned to strength training, aerobic training or a combined strength and aerobic training group. Participants in the exercise group will attend exercise sessions over the course of 9 months at the YMCA. Participants will have opportunities to engage in other activities such as educational run-in visits that will allow for measurement of hemoglobin A1c and emphasize the importance of exercise in improving Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Recent hemoglobin A1c result between 6.5%-13%
* Diagnosis of Type 2 Diabetes Mellitus
* BMI between 18.5 -25 kg/m2
* Blood pressure < 160/100
* Sedentary lifestyle
* Able and willing to enroll and meet requirements of the study

Exclusion Criteria:

* Age less than 30 years or greater than 75 years
* Type 1 diabetes or use of insulin pump
* Triglycerides >500 mg/dL
* Use of weight loss medication
* Bariatric surgery
* Consumes >14 alcoholic drinks per week
* Pregnancy
* Plans to be away for more than four weeks
* Medical conditions which would prevent long-term participation or which would contraindicate physical activity

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2016-02; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c across study visits | Baseline, monthly (for 9 months), 9-Months

SECONDARY OUTCOMES:
Change in body composition across study visits, as measured using DEXA | Baseline, 9-Months
Change in waist circumference across study visits | Baseline, 9-Months
Change in blood pressure across study visits | Baseline, 9-Months
Change in body weight across study visits | Baseline, 9-Months
Changes in cardiorespiratory fitness, as measured by 6-minute walk test | Baseline, 9-Months
Change in muscle strength and endurance, as measured by Biodex strength testing | Baseline, 9-Months
Change in quality of life | Baseline, 9-Months
Change in Dietary Intake, as measured by Food Frequency Questionnaire | Baseline, 9-Months

CONTACTS AND LOCATIONS:
Overall Officials: Latha Palaniappan, MD, MS, Principal Investigator — Stanford School of Medicine
Locations (1):
- Stanford, Palo Alto, California, United States

REFERENCES:
- [Background] Faroqi L, Bonde S, Goni DT, Wong CW, Wong M, Walai K, Araya S, Azamey S, Schreiner G, Bandy M, Raghuram SS, Mittal A, Mukherji A, Wangdak T, Talamoa R, Vera K, Nacif-Coelho C, Cde LG, Christensen M, Johannsen N, Haddad F, Moharir M, Palaniappan L. STRONG-D: Strength training regimen for normal weight diabetics: Rationale and design. Contemp Clin Trials. 2019 Mar;78:101-106. doi: 10.1016/j.cct.2019.01.005. Epub 2019 Jan 6. PMID 30625372
- [Derived] Kobayashi Y, Long J, Dan S, Johannsen NM, Talamoa R, Raghuram S, Chung S, Kent K, Basina M, Lamendola C, Haddad F, Leonard MB, Church TS, Palaniappan L. Strength training is more effective than aerobic exercise for improving glycaemic control and body composition in people with normal-weight type 2 diabetes: a randomised controlled trial. Diabetologia. 2023 Oct;66(10):1897-1907. doi: 10.1007/s00125-023-05958-9. Epub 2023 Jul 26. PMID 37493759